CLINICAL TRIAL: NCT03815669
Title: Improving Quality of Treatment for Shoulder Patients
Status: Terminated | Type: Observational
Why Stopped: Due to covid 19, it has not been possible to recruit enough participants to complete the study.
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: LSskulder
Record Dates: First submitted 2019-01-22; First posted 2019-01-24 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2019-01

CONDITIONS: Arthroscopic Subacromial Decompression
Keywords: arthroscopic subacromial decompression; shoulder impingement syndrome; effect; surgery
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arthroscopic subacromial decompression: Patients referred to arthroscopic subacromial decompression
  Interventions: Procedure: Arthroscopic subacromial decompression

INTERVENTIONS:
Procedure: Arthroscopic subacromial decompression — Arthroscopic subacromial decompression

SUMMARY:
Introduction:

Previous studies indicate that patient characteristics and clinical and psychological factors are related to the effect of surgical treatment but more knowledge about predictors is important in the selection of patients for arthroscopic subacromial decompression.

Objective:

To identify patient characteristics and clinical and psychological factors for pre-operatively predicting the effect of arthroscopic subacromial decompression.

Method:

Patients meting the inclusion criteria will consecutively be enrolled in the study when referred to arthroscopic subacromial decompression. Prior to surgery, patient characteristics and clinical data will be collected. At six and twelve month postoperatively, the effect of the surgical treatment will be assessed. The relationship between effect of surgery and patient characteristics and clinical factors collected at baseline will be examined.

DETAILED DESCRIPTION:
Introduction: Shoulder disorders are the third most common musculoskeletal reason for seeking medical care and accounts for approximately 1% of all visits to the general practitioner and for up to 10% of all referrals to physiotherapists. The prevalence of shoulder disorders has been reported to range from 7% to 26% with some indication that the prevalence increases with age. Subacromial impingement syndrome (SIS) is usually described as a symptomatic irritation of the rotator cuff and the subacromial bursa, and it is considered as one of the most common shoulder disorders. Patients with SIS may present symptoms such as pain during activity, pain at night, loss of muscle strength, and stiffness. Because the shoulder stabilizes the upper limb in its activities, these symptoms affect the performance of tasks essential to daily living. Shoulder disorders produce significant impairments in function and health related quality of life (HR-QoL), and results in substantial health care utilization. SIS frequently affects the working population and is an important cause of sick leave.

Treatment of SIS consists of either conservative- or surgical treatment. Conservative treatments include rest, physiotherapy, non-steroid anti inflammatory drugs (NSAID) and glucocorticoid injections, while surgical treatment consists of arthroscopic or open subacromial decompression, bursectomy and rotator cuff repair. Physiotherapy interventions are recommended as first choice of treatment, while surgical treatment can be considered for those who fail to respond to conservative treatment after 3-6 months. Several studies comparing the effect of arthroscopic subacromial decompression (ASAD) and supervised physiotherapy exercises, have found no significant differences in outcomes between the two treatment strategies.

In Denmark, the number of patients with SIS has increased by 36% from 2006 to 2010. The number of patients treated surgically has increased by 60% to approximately 6500 a year in the same period. Similar increases are reported in other countries.

The literature indicates that some patients do not benefit from ASAD, and success rates between 65-80% have been reported. In Denmark, 10% of employed patients retire prematurely within two years after surgery. Results of studies investigating if ASAD is more effective in selected subgroups of patients showed that clinical and radiological factors and patient characteristics such as sociodemographic, duration of symptoms and duration of sick leave, were associated with the effect of treatment. In addition, psychological factors are reported to impact outcome in both shoulder patients, and other orthopaedic patients. A preoperative scoring system to select patients for ASAD has been developed. However, this focuses on clinical and radiographic factors, and does not consider patient characteristics and psychological factors. Knowledge about predictors for the effect of ASAD in a broader perspective will be of great importance, from both a patient- and an economic perspective.

Aim: The overall aim of the study is to identify patient characteristic and clinical and psychological factors that preoperatively can predict which patients will achieve effect of ASAD. Furthermore, to investigate the quality of objective methods to assess shoulder function, and the association between patient reported outcome measures (PROMs) and objective outcome measures.

Power considerations: Based on data extracted from the Central Denmark Region Electronic Patient Journal (Mid EPJ) an estimation of 150 patients annually undergo ASAD at Aarhus University Hospital. With a planned inclusion period of two years and a drop out rate of 10%, it means that 270 patients will be included. Using an estimate of 20% it is expected that 54 out of 270 patients will not benefit from ASAD. The number of patients without the effect of ASAD will affect the number of potential predictors that can be analyzed.

Outcome assessment: Effect of surgical treatment will be assessed with two instruments: 1) patient evaluated success of treatment with the response options: much improved, moderate improved, unchanged, moderate worse, and much worse and 2) the Oxford Shoulder Score (OSS). Effect of surgical treatment will be defined as a much - or moderate improvement evaluated by the patient, or an improvement of more than 12 points in OSS between baseline and follow-up. The 12 point criterion is previous used to develop a preoperative scoring system to select patients for ASAD.

ELIGIBILITY:
Inclusion Criteria:

* treated with arthroscopic subacromial decompression

Exclusion Criteria:

* Frozen shoulder, full-thickness tear, osteoarthritis, trauma, cancer or neurologic disorders
* Previous surgical treatment in the affected shoulder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients from Department of Orthopaedic Surgery, Aarhus University Hospital, Denmark will consecutively be invited to participate in the study when they are referred to arthroscopic subacromial decompression.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Treatment effect | 12 month postoperatively
  Patient evaluated success of treatment, 5 point Likert scale, Posible answers: much improved, moderate improved, unchanged, moderate worse, much worse
Function | Baseline
  Questionnaire, Oxford Shoulder Score (OSS) 12 questions, each rated on a 5 point Likert scale from 1 to 5, total sum score reported, minimum score 12, maximun score 60, higher scores represent worst outcome
Function | 12 month postoperatively
  Questionnaire, Oxford Shoulder Score (OSS) 12 questions, each rated on a 5 point Likert scale from 1 to 5, total sum score reported, minimum score 12, maximun score 60, higher scores represent worst outcome
Pain self-efficacy | Baseline
  Questionnaire, Pain Self-Efficacy Questionnaire 10 questions, each question rated on a 7-point numeric rating scale from 0 to 6, total sum score reported, minimum score 0, maximun score 60, higher scores indicate greater self-efficacy
Pain self-efficacy | 12 month postoperatively
  Questionnaire, Pain Self-Efficacy Questionnaire 10 questions, each question rated on a 7-point numeric rating scale from 0 to 6, total sum score reported, minimum score 0, maximun score 60, higher scores indicate greater self-efficacy
Health related quality of life | Baseline
  Questionnaire, EQ-5D-5L 5 questions representing 5 dimentions, each question rated on a 5-point Likert scale from 1 to 5, higher scores indicate worse outcome, EQ VAS scale representing overall Health status, rated from 0 to 100, higher score indicate better outcome
Health related quality of life | 12 month postoperatively
  Questionnaire, EQ-5D-5L 5 questions representing 5 dimentions, each question rated on a 5-point Likert scale from 1 to 5, higher scores indicate worse outcome, EQ VAS scale representing overall Health status, rated from 0 to 100, higher score indicate better outcome
Anxiety and depression | Baseline
  Questionnaire, Hospital Anxiety and Depression Scale (HADS) 14 questions, 7 questions related to the subscale Anxiety, 7 questiion related to the subscale Depression, each question rated on a 4-point Likert scale from 0 to 3, total sum score for each subscale reported, higher scores indicate worse outcome
Anxiety and depression | 12 month postoperatively
  Questionnaire, Hospital Anxiety and Depression Scale (HADS) 14 questions, 7 questions related to the subscale Anxiety, 7 questiion related to the subscale Depression, each question rated on a 4-point Likert scale from 0 to 3, total sum score for each subscale reported, higher scores indicate worse outcome
Fear-Avoidance beliefs | Baseline
  Questionnaire, Fear-Avoidance Beliefs Questionnaire (FABQ) 16 items, 4 items related to the physical activity subscale, 7 items related to the Work subscale, 5 items not used in the scoring, each item rated on a 7-point Likert scale from 0 to 6, total sumscore for each subscale reported, minimum scores 0, maximum scores for the physical activity subscale 24, maximal score for the Work subscale 42, higher scores indicate worse outcome
Fear-Avoidance beliefs | 12 month postoperatively
  Questionnaire, Fear-Avoidance Beliefs Questionnaire (FABQ) 16 items, 4 items related to the physical activity subscale, 7 items related to the Work subscale, 5 items not used in the scoring, each item rated on a 7-point Likert scale from 0 to 6, total sumscore for each subscale reported, minimum scores 0, maximum scores for the physical activity subscale 24, maximal score for the Work subscale 42, higher scores indicate worse outcome
Pain, VAS | Baseline
  Pain at rest, activity and at night, Visual Analogue Scale (VAS) Scale rating form 0 to 10, higher score indicate worse outcome
Pain, VAS | 6 month postoperatively
  Pain at rest, activity and at night, Visual Analogue Scale (VAS) Scale rating form 0 to 10, higher score indicate worse outcome
Muscle strength | Baseline
  Internal and external rotation, abduction
Muscle strength | 6 month postoperatively
  Internal and external rotation, abduction
Range of motion (ROM) | Baseline
  Internal and external rotation, abduction and flexion
Range of motion (ROM) | 6 month postoperatively
  Internal and external rotation, abduction and flexion
Motor and process skills | Baseline
  The Assessment of Motor and Process Skills (AMPS)
Motor and process skills | 6 month postoperatively
  The Assessment of Motor and Process Skills (AMPS)
Return to work | Baseline
  Duration of sick leave
Comorbidity | Baseline
  Charlson comorbidity index

SECONDARY OUTCOMES:
Treatment effect | 6 month postoperatively
  Patient evaluated success of treatment, 5 point Likert scale, Posible answers: much improved, moderate improved, unchanged, moderate worse, much worse
Function | 6 month postoperatively
  Questionnaire, Oxford Shoulder Score (OSS) 12 questions, each rated on a 5 point Likert scale from 1 to 5, total sum score reported, minimum score 12, maximun score 60, higher scores represent worst outcome
Pain self-efficacy | 6 month postoperatively
  Questionnaire, Pain Self-Efficacy Questionnaire 10 questions, each question rated on a 7-point numeric rating scale from 0 to 6, total sum score reported, minimum score 0, maximun score 60, higher scores indicate greater self-efficacy
Health related quality of life | 6 month postoperatively
  Questionnaire, EQ-5D-5L 5 questions representing 5 dimentions, each question rated on a 5-point Likert scale from 1 to 5, higher scores indicate worse outcome, EQ VAS scale representing overall Health status, rated from 0 to 100, higher score indicate better outcome
Anxiety and depression | 6 month postoperatively
  Questionnaire, Hospital Anxiety and Depression Scale (HADS) 14 questions, 7 questions related to the subscale Anxiety, 7 questiion related to the subscale Depression, each question rated on a 4-point Likert scale from 0 to 3, total sum score for each subscale reported, higher scores indicate worse outcome
Fear-Avoidance beliefs | 6 month postoperatively
  Questionnaire, Fear-Avoidance Beliefs Questionnaire (FABQ) 16 items, 4 items related to the physical activity subscale, 7 items related to the Work subscale, 5 items not used in the scoring, each item rated on a 7-point Likert scale from 0 to 6, total sumscore for each subscale reported, minimum scores 0, maximum scores for the physical activity subscale 24, maximal score for the Work subscale 42, higher scores indicate worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Annemette Krintel Petersen, Ph.D, Study Director — Dept. of Clinical Medicine, Aaarhus University
Locations (1):
- Dept of Orthopaedic Surgery and dept. of Physiotherapy and Occupational Therapy, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided